CLINICAL TRIAL: NCT06367595
Title: Effect of Intrathecal Magnesium Sulfate Versus Intravenous Magnesium Sulfate on Postoperative Pain After Abdominal Hysterectomy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Salah Hassanein, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Intrathecal MgSO4
Record Dates: First submitted 2024-02-20; First posted 2024-04-16 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Abdominal Hysterectomy
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- intrathecal (Active Comparator): will include 30 patients who will receive
  * Intrathecal hyperbaric bupivacaine 0.5 % 20 mg in 4 ml plus magnesium sulfate 30 mg of 0.5 ml volume.
  * 250 ml of isotonic saline infusion over 15 minutes immediately before spinal anesthesia, then 250 ml of isotonic saline infusion over 2 hours.
  Interventions: Drug: Magnesium sulfate
- intravenous (Active Comparator): will include 30 patients who will receive
  - 30 mg/kg magnesium sulfate at a concentration of 100 mg/ml (regarding the ideal body weight) in 250 ml of isotonic saline infusion over 15 minutes immediately before spinal anesthesia (intrathecal hyperbaric bupivacaine 0.5 % 20 mg in 4 ml plus 0.5 ml of isotonic saline), and then 10 mg/kg/h magnesium sulfate in 250 ml isotonic saline infusion over 2 hours.
  Interventions: Drug: Magnesium sulfate
- placebo (Placebo Comparator): will include 30 patients who will receive
  * intrathecal hyperbaric bupivacaine 0.5 % 20 mg in 4 ml plus 0.5 ml of isotonic saline.
  * 250 ml of isotonic saline infusion over 15 minutes immediately before spinal anesthesia then 250 ml of isotonic saline infusion over 2 hours.
  Interventions: Drug: Magnesium sulfate

INTERVENTIONS:
Drug: Magnesium sulfate — IV magnesium sulfate versus magnesium sulfate to intrathecal hyperbaric bupivacaine

SUMMARY:
The present study aims to compare the effect of adding IV magnesium sulfate versus magnesium sulfate to intrathecal hyperbaric bupivacaine in total abdominal hysterectomy regarding the duration of postoperative analgesia, hemodynamic stability, and complications.

DETAILED DESCRIPTION:
Abdominal Hysterectomy (AH) is associated with an intense inflammatory response that can result in moderate to severe postoperative pain, sometimes difficult to control.

Postoperative pain can cause many complications such as restlessness, increased sympathetic activity, high blood pressure, and tachycardia. Opioids are effective analgesics; however, they produce unwanted side effects, such as respiratory depression, nausea, and vomiting. Nonopioid drugs can decrease opioid usage and dependency.

Different adjuvants have been added to local anesthetics to increase the duration of the regional anesthesia, decrease pain-relieving drugs, and delay the onset of postoperative pain.

According to numerous reports, Magnesium sulfate has analgesic effects and lowers opioid consumption in many surgeries especially abdominal surgeries.

The analgesic properties of magnesium are based on acting as a non-competitive antagonist of N-Methyl-D-Aspartate (NMDA) receptors in central nervous system and regulating the calcium influx into the cell. These properties avoid the central sensitization mechanisms due to the stimulation of peripheral nociceptive nerves In the spinal cord, magnesium sulfate decreases pain transmission by hyperpolarizing spinal interneurons via G-protein-mediated activation of potassium channels and by decreasing the release of the neurotransmitters (substance P and glutamate) from primary afferent terminals.

Adequate postoperative pain relief can enhance recovery and increase patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 40-65 years old
* Patients with ASA clinical status I/II
* Patients eligible for abdominal hysterectomy
* Oncological surgery

Exclusion Criteria:

* Body mass index (BMI) ≥ 40/kg / m2
* Previous abdominal surgery (except cesarean section)
* Severe cardiovascular, renal, and hepatic dysfunction
* Contraindications to spinal anesthesia
* Neuromuscular diseases
* Inappropriate for spinal anesthesia
* Patient refusal

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
effect on postoperative pain after abdominal hysterectomy using visual analog score | Baseline
  the pain intensity assessment at rest and on movement (from lying to sitting on the bed) using Visual analog score (VAS) This will measure pain intensity from 0 to 10 (goal is to be < 4) 0: no pain 3: mild pain 7: moderate pain 10: severe pain

SECONDARY OUTCOMES:
sedation by Ramsay sedation scale | Baseline
  From 1 to 6
  1. Patient is anxious and agitated or restless, or both.
  2. Patient is cooperative, oriented, and tranquil.
  3. Patient responds to commands only.
  4. Patient exhibits brisk response to light glabellar tab or loud auditory stimulus.
  5. Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus.
  6. Patient exhibits no response.
time of the first opioid request | Baseline
  time of the first opioid request, concentration and the occurrence of complications (hypotension, bradycardia, itching, urinary retention.) all over 24 hours postoperatively.
Mean arterial blood pressures (MAP) | Baseline
  mean arterial blood pressures (MAP) will be recorded at time 0 then every 15 minutes in the first 2 hours, then at 6, 12, 24 hours postoperatively.
Heart rate (HR) | Baseline
  Heart rate (HR) will be recorded at time 0 then every 15 minutes in the first 2 hours, then at 6, 12, 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy A Youssef, Professor, Study Chair — Assuit University Hospital; Mohamed F Mostafa, Ass professor, Study Chair — Assuit University Hospital; Ahmed M Elsonbaty, Lecturer, Study Director — Assuit University Hospital; Marwa S Hassanein, Resident, Principal Investigator — Assuit University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brandsborg B. Pain following hysterectomy: epidemiological and clinical aspects. Dan Med J. 2012 Jan;59(1):B4374. PMID 22239844
- [Background] Kim TK, Yoon JR. Comparison of the neuroendocrine and inflammatory responses after laparoscopic and abdominal hysterectomy. Korean J Anesthesiol. 2010 Oct;59(4):265-9. doi: 10.4097/kjae.2010.59.4.265. Epub 2010 Oct 21. PMID 21057617
- [Background] Wu CL, Fleisher LA. Outcomes research in regional anesthesia and analgesia. Anesth Analg. 2000 Nov;91(5):1232-42. doi: 10.1097/00000539-200011000-00035. No abstract available. PMID 11049915
- [Background] Camu F, Van Aken H, Bovill JG. Postoperative analgesic effects of three demand-dose sizes of fentanyl administered by patient-controlled analgesia. Anesth Analg. 1998 Oct;87(4):890-5. doi: 10.1097/00000539-199810000-00027. PMID 9768789
- [Background] Koltka K, Uludag E, Senturk M, Yavru A, Karadeniz M, Sengul T, Ozyalcin S. Comparison of equipotent doses of ropivacaine-fentanyl and bupivacaine-fentanyl in spinal anaesthesia for lower abdominal surgery. Anaesth Intensive Care. 2009 Nov;37(6):923-8. doi: 10.1177/0310057X0903700606. PMID 20014598
- [Background] Buvanendran A, McCarthy RJ, Kroin JS, Leong W, Perry P, Tuman KJ. Intrathecal magnesium prolongs fentanyl analgesia: a prospective, randomized, controlled trial. Anesth Analg. 2002 Sep;95(3):661-6, table of contents. doi: 10.1097/00000539-200209000-00031. PMID 12198056
- [Background] De Oliveira GS Jr, Castro-Alves LJ, Khan JH, McCarthy RJ. Perioperative systemic magnesium to minimize postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2013 Jul;119(1):178-90. doi: 10.1097/ALN.0b013e318297630d. PMID 23669270
- [Background] Do SH. Magnesium: a versatile drug for anesthesiologists. Korean J Anesthesiol. 2013 Jul;65(1):4-8. doi: 10.4097/kjae.2013.65.1.4. Epub 2013 Jul 19. PMID 23904932
- [Background] Ishii H, Kohno T, Yamakura T, Ikoma M, Baba H. Action of dexmedetomidine on the substantia gelatinosa neurons of the rat spinal cord. Eur J Neurosci. 2008 Jun;27(12):3182-90. doi: 10.1111/j.1460-9568.2008.06260.x. Epub 2008 Jun 1. PMID 18554299
- [Background] Shang AB, Gan TJ. Optimising postoperative pain management in the ambulatory patient. Drugs. 2003;63(9):855-67. doi: 10.2165/00003495-200363090-00002. PMID 12678572
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382
- [Background] Khan BA, Guzman O, Campbell NL, Walroth T, Tricker JL, Hui SL, Perkins A, Zawahiri M, Buckley JD, Farber MO, Ely EW, Boustani MA. Comparison and agreement between the Richmond Agitation-Sedation Scale and the Riker Sedation-Agitation Scale in evaluating patients' eligibility for delirium assessment in the ICU. Chest. 2012 Jul;142(1):48-54. doi: 10.1378/chest.11-2100. PMID 22539644
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Yazdi AP, Esmaeeli M, Gilani MT. Effect of intravenous magnesium on postoperative pain control for major abdominal surgery: a randomized double-blinded study. Anesth Pain Med (Seoul). 2022 Jul;17(3):280-285. doi: 10.17085/apm.22156. Epub 2022 Jul 28. PMID 35918860
- [Background] Benevides ML, Fialho DC, Linck D, Oliveira AL, Ramalho DHV, Benevides MM. Intravenous magnesium sulfate for postoperative analgesia after abdominal hysterectomy under spinal anesthesia: a randomized, double-blind trial. Braz J Anesthesiol. 2021 Sep-Oct;71(5):498-504. doi: 10.1016/j.bjane.2021.01.008. Epub 2021 Mar 21. PMID 33762190